CLINICAL TRIAL: NCT02478788
Title: Neuroimaging Study of Risk Factors for Adolescent Bipolar Disorder
Acronym: NERF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Melissa Delbello, Academic Medical Director, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: DelBello/McNamara Neuroimaging; R01MH097818-01A1 (NIH)
Record Dates: First submitted 2015-06-15; First posted 2015-06-23 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- LR-MAS - Low-risk ADHD adolescents (Experimental): ADHD adolescents without any first or second degree-relatives with bipolar disorder. Low-risk ADHD adolescents (n=60) will receive treatment with open-label mixed amphetamine salts-extended release (MAS-XR), which is approved by the United States Food and Drug Administration (USFDA) for the treatment of ADHD and is a commonly prescribed psychostimulant medication for adolescents with ADHD.
  Interventions: Drug: mixed amphetamine salts-extended release (MAS-XR)
- HR-MAS - High-risk ADHD adolescents (Experimental): ADHD adolescents with a parent with bipolar disorder ("high-risk"). High-risk ADHD adolescents will be randomized to double-blind treatment with MAS-XR (n=60) or placebo (n=60). The subjects in this group will receive mixed amphetamine salts-extended release( MAS-XR), which is approved by the United States Food and Drug Administration (USFDA) for the treatment of ADHD and is a commonly prescribed psychostimulant medication for adolescents with ADHD.
  Interventions: Drug: mixed amphetamine salts-extended release (MAS-XR)
- HR-P - High-risk ADHD on Placebo (Placebo Comparator): ADHD adolescents with a parent with bipolar disorder ("high-risk"). High-risk ADHD adolescents will be randomized to double-blind treatment with MAS-XR (n=60) or placebo (n=60). Following initiation of treatment, the ADHD adolescents will have regularly scheduled visits during which symptom and tolerability ratings will be performed.
  Interventions: Drug: Placebo
- HC (Healthy Controls) (No Intervention): Healthy subjects (n=60) will be recruited from the community and will not receive medication but will undergo MR scans at the same intervals to assess normal variability in imaging parameters between time points as well as to adjust and interpret comparisons within patients (i.e., whether patient values are changing toward or away from those of healthy adolescents). Neuroimaging evaluations will be performed at baseline and Week 12 (or termination).

INTERVENTIONS:
Drug: mixed amphetamine salts-extended release (MAS-XR) — MAS-XR is a psychostimulant medication composed of amphetamine and dextroamphetamine, has been systematically studied in adolescents with ADHD, and is FDA-approved for the treatment of ADHD in adolescents.
  Other Names: AdderallXR
  Arms: HR-MAS - High-risk ADHD adolescents; LR-MAS - Low-risk ADHD adolescents
Drug: Placebo — Pills with no medication in it
  Arms: HR-P - High-risk ADHD on Placebo

SUMMARY:
The main purpose of this study is to see the affects of the study medication called mixed amphetamine salts-extended release (MAS-XR) on brain function by taking brain pictures. The researchers also want to see if MAS-XR makes your child more or less likely to develop problems like acting out (i.e. periods of irritability, agitation, aggression).

MAS-XR is approved by the United States Food and Drug Administration (FDA) to treat attention deficit hyperactivity disorder (ADHD) in adults, children and adolescents.

DETAILED DESCRIPTION:
A 12-week prospective study of two groups of adolescents (ages 10-18 years) with attention deficit/hyperactivity disorder (ADHD); 1) ADHD adolescents with a first degree relative with bipolar disorder ("high-risk") and 2) ADHD adolescents without any first or second degree-relatives with a mood disorder ("low-risk"). Patients will be evaluated using diagnostic interviews and symptom ratings, will receive neuroimaging scans (fMRI, DTI, 1H MRS), and will then be assigned to treatment. Low-risk ADHD adolescents (n=60) will receive treatment with open-label mixed amphetamine salts-extended release (MAS-XR), which is approved by the United States Food and Drug Administration (USFDA) for the treatment of ADHD and is a commonly prescribed psychostimulant medication for adolescents with ADHD. High-risk ADHD adolescents will be randomized to double-blind treatment with MAS-XR (n=60) or placebo (n=60). Following initiation of treatment, the ADHD adolescents will have regularly scheduled visits during which symptom and tolerability ratings will be performed. Healthy subjects (n=60) will be recruited from the community and will not receive medication but will undergo magnetic resonance imaging (MRI) scans at the same intervals to assess normal variability in imaging parameters between time points as well as to adjust and interpret comparisons within patients (i.e., whether patient values are changing toward or away from those of healthy adolescents). Neuroimaging (fMRI, DTI,1H MRS) evaluations will be performed at baseline and Week 12 (or termination).

ELIGIBILITY:
Inclusion Criteria:

* Ages 10-18years old
* If female, not pregnant
* Fluent in English
* No contraindication to an MRI scan (e.g., braces or claustrophobia)
* An IQ > 80
* No unstable or major medical or neurological illness
* No lifetime DSM-5 substance use disorder
* Lives <100 miles from the University of Cincinnati
* Provision of written informed consent/assent
* At least one biological first degree relative with bipolar I disorder ('high-risk' only)
* No first- or second-degree relative with a mood or psychotic disorder ('low-risk' and healthy controls only) with the exception of late onset depressive disorders.
* No lifetime DSM-5 Axis I disorder (other than specific phobias, healthy controls only).
* No medications with CNS effects within 5 half-lives from baseline MR scan (healthy controls only).

Inclusion criteria for 'high-risk' and 'low-risk' ADHD subjects :

* Meets DSM-5 criteria for ADHD, inattentive, hyperactive/impulsive, or combined type
* No exposure to psychostimulants or ADHD medications in the 3 months prior to baseline
* No lifetime exposure to mood stabilizers or antipsychotic medications
* No concomitant use of any psychotropic medication other than study medications during study participation
* No history of intolerance, hypersensitivity, or non-response to MAS-XR
* No comorbid mood, anxiety, conduct, eating or psychotic disorder that in the opinion of the primary investigator is the current and primary focus of treatment. No Tourette's disorder, chronic tic disorder, or autism spectrum disorder.
* No clinically significant ECG or blood pressure abnormalities
* No family history of sudden death or ventricular arrhythmia

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 153 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Baseline-endpoint change in prefrontal-amygdala functional connectivity by fMRI. | Baseline and up to 12 weeks
  Using functional magnetic resonance imaging (fMRI), change in prefrontal-amygdala functional connectivity will be determined by contrasting baseline and endpoint blood oxygen level-dependent (BOLD) activity in the amygdala and prefrontal cortex (BA47) during performance of the CPT-END task, and determining the prefrontal-amygdala interrelationship using a seed-region (amygdala) based functional connectivity analysis.

SECONDARY OUTCOMES:
Baseline-endpoint change in uncinate fasciculus white matter integrity by DTI | Baseline and up to 12 weeks
  Change in uncinate fasciculus white matter integrity will be determined by contrasting baseline and endpoint fractional anisotropy using diffusion tensor imaging (DTI).
Baseline-endpoint change in glutamate (Glu) and N-acetyl aspartate (NAA) concentrations in the prefrontal cortex (BA47) by 1H MRS. | Baseline and up to 12 weeks
  This is a composite measure of change in right and left prefrontal cortex (BA47) Glu and NAA concentrations (mM). It will be determined by contrasting baseline and endpoint levels using proton magnetic resonance spectroscopy (1H MRS).

CONTACTS AND LOCATIONS:
Overall Officials: Robert McNamara, PhD, Study Director — University of Cincinnati
Locations (1):
- University of Cincinnati, Department of Psychiatry and Behavioral Neuroscience, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Qin K, Pan N, Lei D, Zhu Z, Tallman MJ, Patino LR, Gong Q, Sweeney JA, DelBello MP, McNamara RK. Different Changes in Brain Functional Networks Following 12-Week Psychostimulant Treatment in Attention-Deficit/Hyperactivity Disorder Youth With and Without Familial Risk for Bipolar I Disorder. J Am Acad Child Adolesc Psychiatry. 2025 Jul 23:S0890-8567(25)00751-8. doi: 10.1016/j.jaac.2025.07.421. Online ahead of print. PMID 40712681